CLINICAL TRIAL: NCT04600479
Title: Study on the Prevalence of Hepatitis C In a psychiatRic Population
Acronym: SaPHIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC20_0022
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; psychiatry; Hepatitis B; HIV; care pathway
MeSH Terms: conditions — Hepatitis C; Hepatitis B

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- prevalence and follow-up of HCV positive patients (Experimental): 1. Cross-sectional assessment of prevalence : evaluation of the prevalence of HCV, HBV and HIV viral infections
  2. Cohort follow-up of HCV positive patients : evaluation of care pathway and barriers to care for hepatitis C
  Interventions: Diagnostic Test: Evaluation of the prevalence of HCV, HBV and HIV viral infections

INTERVENTIONS:
Diagnostic Test: Evaluation of the prevalence of HCV, HBV and HIV viral infections — 1. Assessment of prevalence HCV, HBV and HIV prevalence estimations. Sociodemographic and clinical data will be collected from the patient's medical record and through self-questionnaires completed by the patient. A systematic screening by 3 RDTs (HCV, HBV and HIV) will be proposed in the specific framework of the SaPHIR study.This is a screening performed on capillary blood (TOYO VHC ®, TOYO VHB ® and INSTI HIV 1 / HIV 2 ®), to obtain a result in less than 30 minutes.
     In case of confirmation of the diagnosis of viral hepatitis or HIV infection, the final result will be transmitted and explained to the patient by the referring doctor, who will organize the adapted care pathway and prescribe the DAA for the simple patients. The complex patients will be referred to the specialist to consider starting an appropriate treatment.
  2. Evaluation of care pathway and barriers to care for hepatitis C. Only patients with positive HCV RDT participating in this follow-up.

SUMMARY:
Viral hepatitis, especially hepatitis C, is a major public health issue. Nowadays, very few studies in France have evaluated the prevalence of hepatitis C in a psychiatric environment.

In 2019, at the time of new treatments for HCV, it therefore seems essential to update the available data by estimating the prevalence of chronic active hepatitis C in psychiatric population. In addition to an update of epidemiological data, it is of high importance to assess the effectiveness of the care pathway for patients in whom chronic active hepatitis C is diagnosed, including the cascade of care, currently too inefficient despite treatments that are themselves ultra-efficient. Indeed, it is essential that once hepatitis is detected, it is formally diagnosed, then that the patient actually starts care and is adherent to treatment (take his treatment according to the prescription and until the end: this implies that the patient accepts his or her illness and understands the value of the prescribed treatments), to hope to cure the infection.

In this context, the SaPHIR study will allow to test a systematic screening of patients in an adult psychiatric environment, through rapid diagnostic tests (RDT). The objective is to promote the adherence of patients, and to assess possible obstacles in order to optimize the screening (RDTs), diagnosis (confirmation of only positive RDTs by venous sampling) and care management circuits in routine practice. In addition, the study envisages a combined HCV-HBV-HIV screening, taking into account the cross-infection risk (same mode of contamination, same risk population, frequent co-infections, more severe liver pathology in case of co-infection, etc.), thus making it possible to take care of the patient as a whole. The results of the SaPHIR study can ultimately be sent to the French health authorities to improve screening and care circuits, and their coverage by social security.

DETAILED DESCRIPTION:
Participation in the SaPHIR study will be offered to patients admitted to one of the inpatient or outpatient adult psychiatric units of the hospitals participating in the study (around Nantes), provided that the realization of the RDTs will be possible.

1. Cross-sectional assessment of prevalence : evaluation of the prevalence of HCV, HBV and HIV viral infections All patients admitted to one of the inpatient or outpatient adult psychiatric units of the hospitals participating in the study, whatever the psychiatric diagnosis and without age limit, may be included in the study, provided that the realization of the RDTs will be possible. Only patients who will accept the realization of the HCV RDT will be included, in order to be able to respond to the primary objective of the study. The agreement to realize the two other RDTs is optional. However, for patients who already had a HCV serology performed less than 3 months before inclusion, the HCV RDT will not be performed and the data collected for the study will be based on the previous serology.
2. Cohort follow-up of HCV positive patients : evaluation of care pathway and barriers to care for hepatitis C Patients who are included in the cross-sectional assessment of prevalence of the SaPHIR study and having a positive HCV RDT (or positive HCV serology performed less than 3 months ago) will participate in the follow-up of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Cross-sectional assessment of prevalence

   Patients with all the following characteristics can be included:
   * Patient admitted to one of the inpatient or outpatient adult psychiatric units of the hospitals participating in the study
   * Patient accepting the realization of the HCV RDT (or patient with positive HCV serology performed less than 3 month ago)
2. Cohort follow-up of HCV positive patients:

Patients who are included in the cross-sectional assessment of prevalence of the SaPHIR study and having a positive HCV RDT (or positive HCV serology performed less than 3 months ago) will participate in the follow-up of the study.

Exclusion Criteria:

1. Cross-sectional assessment of prevalence:

   Patients with at least one of the following characteristics cannot be included:
   * Minors under 15 years of age (all units involved in the recruitment are adult psychiatry units, for which the minimum age limit is 15 years and 3 months);
   * Pregnant or lactating woman;
   * Participating simultaneously in another interventional research on a drug (so as not to interfere with the biological assays);
   * Not mastering the reading and writing of the French language well enough.
   * Patient placed under judicial protection
2. Cohort follow-up of HCV positive patients Patients who are included in the cross-sectional assessment of prevalence of the SaPHIR study, with negative RDT HCV (or negative HCV serology performed less than 3 months ago) cannot participate in the follow-up of the study.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 796 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Estimation of the prevalence of chronic hepatitis C in a psychiatric population | 33 months
  The prevalence estimate will be based on the percentage of patients in whom the viral C RNA is detected (greater than 15 IU / mL) in venous blood by the polymerase chain reaction (PCR) technique, among the patients admitted to one of the inpatient or outpatient adult psychiatric units of the hospitals participating in the study (around Nantes). The viral C RNA will be considered undetected in the case of a negative HCV RDT screening.

SECONDARY OUTCOMES:
Effectiveness of the care pathway of the HCV-infected patient | 33 months
  Percentage of patients who accepted the RDT screening Percentage of patients screened positive Percentage of patients who accepted venous sampling to achieve the C viral load Percentage of patients diagnosed positive by carrying out the C viral load Percentage of patients (diagnosed as positive) having started a care procedure Percentage of patients referred to specialists Percentage of compliant patients Percentage of patients considered cured 12 weeks after the end of treatment
Prevalence of hepatitis C in a psychiatric population (cured hepatitis and chronic active hepatitis) | 33 months
  The estimate of the prevalence of hepatitis C will be based on the percentage of patients with positive screening by RDT (anti-HCV Ab), among all the patients included in the study.
Prevalence of active hepatitis B in a psychiatric population | 33 months
  The estimate of the prevalence of active hepatitis B will be based on the percentage of patients with positive screening by RDT (HBs Ag), among all patients included in the study. The percentage of patients with a confirmation of the diagnosis of hepatitis B by B viral load (PCR) on venous blood will also be documented.
Prevalence of HIV in a psychiatric population | 33 months
  The estimate of the prevalence of HIV infection will be based on the percentage of patients screened by RDT (recombinant proteins gp41 / gp 46), among all patients included in the study. The percentage of patients with a confirmation of the diagnosis of HIV infection by HIV screening (combined anti-HIV1, anti-HIV2 and anti-HIV P24 (HIV1)) on venous blood will also be documented.
Prevalence of HCV-HBV-HIV co-infections in a psychiatric population | 33 months
  The estimate of the prevalence of HIV-HCV-HBV co-infections will be based on the percentages of patients co-infected with VHC-VHB, VHC-VIH, VIH-VHB or VHC-VHB-VIH, among all patients included in the study.
Prevalence of hepatitis C in the sub-population of IDU patients | 33 months
  The estimate of the prevalence of hepatitis C in the sub-population of IDU will be based on the percentages of IDU patients with positive screening by RDT (anti-HCV ab), among all the patients included in the study.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHS de Blain, Blain
  - CH Georges Daumézon, Bouguenais
  - CHU Nantes, Nantes